CLINICAL TRIAL: NCT05501379
Title: Comparison of the Physical Activity Assessed by an Accelerometer and the International Physical Activity Questionnaire in Oncologic Patients
Brief Title: Comparison of the Physical Activity in Cancer Patients Assessed by Questionnaire and Motion Tracker
Acronym: OncoPhys
Status: Recruiting | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 067/22
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma; Pancreas Cancer; Colorectal Cancer
Keywords: Physical Activity; Accelerometer; International Physical Activity Questionnaire; Cancer Therapy; GeneActiv; Quality of Life; Fatigue
MeSH Terms: conditions — Lymphoma; Pancreatic Neoplasms; Colorectal Neoplasms; Motor Activity; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients: Patients with a verified diagnosis of lymphoma, colorectal or pancreatic cancer requiring surgical, chemo or radio therapy.
  Interventions: Other: No intervention - observational study only

INTERVENTIONS:
Other: No intervention - observational study only — No intervention - observational study only

SUMMARY:
Physical activity is an important aspect of cancer therapy but correct measurement of physical activity is difficult. In this study, the physical activity of patients undergoing cancer therapy is assessed by questionnaire and by motion tracker. The results are then compared to answer whether there are differences between the two measurements. Findings of this study will help to improve the assessment of physical activity in cancer patients.

DETAILED DESCRIPTION:
Although physical activity has been identified as a relevant determinant of cancer therapy outcome, its valid assessment remains challenging. In principle, direct and indirect assessment instruments can be employed for assessment of physical activity. While direct instruments, e.g. accelerometers, are considered to provide a more objective measurement, indirect tools such as questionnaires are less expensive and more applicable for use in larger study populations. The validity of both forms of measurements in cancer patients is however not well studied. Therefore, this study aims to elucidate the relative validity of an accelerometer in comparison to a standardized physical questionnaire at different time points of cancer therapy. Findings of this study will allow conclusions regarding the ideal modalities for assessment of physical activity in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* verified diagnosis of lymphoma, colorectal or pancreatic cancer
* requirement of surgical, chemo or radio therapy
* provision of informed consent

Exclusion Criteria:

* pregnancy
* inability to provide consent
* use of a rollator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at University Medicine Greifswald (Northeast Germany). Patients with the verified diagnosis of lymphoma, colerectal or pancreatic cancer requiring surgical, chemo or radio therapy will be identified in the respective wards or day care units of the hosptial.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of physical activity assessments within 1 week after initiation of cancer therapy | 1 week after initiation of cancer therapy
  Difference in physical activity measured by the GeneActiv accelerometer and the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)

SECONDARY OUTCOMES:
Comparison of physical activity assessments 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Difference in physical activity measured by the GeneActiv accelerometer and the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Comparison of changes in physical activity between assessements within 1 week and 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Difference in changes of physical activity measured by the GeneActiv accelerometer and the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of Eastern Co-operative Oncology Group (ECOG) Performance Status to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between ECOG Performance Status and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of Eastern Co-operative Oncology Group (ECOG) Performance Status to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between ECOG Performance Status and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of Karnofsky Performance Status (KPS) to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between KPS and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of Karnofsky Performance Status (KPS) to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between KPS and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of age to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy
  Association between age and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of age to physical activity assessed by questionnaire | 1 week after initiation of cancer therapy
  Association between age and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of sex to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy
  Association between sex and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of sex to physical activity assessed by questionnaire | 1 week after initiation of cancer therapy
  Association between sex and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of quality of life to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between quality of life assessed by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ C-30) and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of quality of life to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between quality of life assessed by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ C-30) and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Therapy-related quality of life | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between quality of life assessed by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ C-30) and cancer therapy modality
Relation of fatigue to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between fatigue assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire (EORTC QLQFA-12) and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of fatigue to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between fatigue assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire (EORTC QLQFA-12) and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Therapy-related fatigue | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between fatigue assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire (EORTC QLQFA-12) and cancer therapy modality
Relation of sleep duration to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep duration measured by the GeneActiv accelerometer in hours and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of sleep duration to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep duration measured by the GeneActiv accelerometer in hours and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of sleep efficiency to physical activity assessed by accelerometer | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep efficiency, i.e. the ratio of sleep duration to total bed time measured by the GeneActiv accelerometer in hours, and physical activity measured by the GeneActiv accelerometer in metabolic equivalents of tasks (METs)
Relation of sleep efficiency to physical activity assessed by questionnaire | 1 week before initiation of cancer therapy, 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep efficiency, i.e. the ratio of sleep duration to total bed time measured by the GeneActiv accelerometer in hours, and physical activity measured by the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Therapy-related sleep duration | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep duration measured by the GeneActiv accelerometer in hours and cancer therapy modality
Therapy-related sleep efficiency | 1 week after initiation of cancer therapy, 12 weeks after initiation of cancer therapy
  Association between sleep efficiency, i.e. the ratio of sleep duration to total bed time measured by the GeneActiv accelerometer in hours, and cancer therapy modality
Changes in fatigue between assessements before and 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Differences in fatigue assessed by the European Organisation for Research and Treatment of Cancer Quality of Life Fatigue Questionnaire (EORTC QLQFA-12)
Changes in quality of life between assessements before and 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Differences in quality of life assessed by the European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ C-30)
Relation of tumor entity to changes in physical activity between assessements within 1 week and 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Association between tumor entity and changes in physical activity measured by the GeneActiv accelerometer and the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)
Relation of cancer therapy modality to changes in physical activity between assessements within 1 week and 12 weeks after initiation of cancer therapy | 12 weeks after initiation of cancer therapy
  Association between cancer therapy modality and changes in physical activity measured by the GeneActiv accelerometer and the short version of the International Physical Activity Questionnaire (IPAQ-sf) in metabolic equivalents of tasks (METs)

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Aghdassi, Professor, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany